CLINICAL TRIAL: NCT00930254
Title: Vascular Ultrasound During the Use of Peripheral Intravenous Catheters in Children: A Clinical, Randomized and Controlled Trial.
Brief Title: Peripheral Intravenous Puncture Guided by Vascular Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Ariane Ferreira Machado Avelar, UNIFESP
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: USV01; 0402/06
Record Dates: First submitted 2009-06-25; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Intravenous Puncture Assertivity; Intravenous Puncture Guided by Vascular Ultrasound; Intravenous Therapy Complications
Keywords: pediatric nursing; peripheral catheterization; ultrasonics; intravenous infusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound (Experimental): Vascular puncture guided by vascular ultrasound
  Interventions: Procedure: IV puncture guided by ultrasound

INTERVENTIONS:
Procedure: IV puncture guided by ultrasound — Comparisons between traditional and ultrasound group
  Other Names: vascular ultrasound

SUMMARY:
This research, aimed to verify whether the use of vascular ultrasonography (VUS) could lead to better results in the peripheral venous access implementation in children.

Objectives: To compare, regardless of the number of venous puncture attempts, peripheral venous access obtained in children, according to VUS use or traditional method for peripheral intravenous catheter (PIC) insertion; assertiveness in the use of PIC in children, defined as success in the first attempt of puncture and PIC withdrawal according to release of treatment, related to VUS or traditional method and to describe the influence of VUS on PIC dwell time and development of local complications related to the use of intravenous therapy in children.

DETAILED DESCRIPTION:
Clinical, randomized and controlled trial, conducted in a pediatric surgery ward of a university hospital in São Paulo. Data collection occurred from February 26th, 2007 to July 07th, 2008, after ethical merits of research approval. The sample comprised 382 venous puncture randomly allocated in the experimental group (EG), venous puncture guided by VUS, or in the control group (CG), traditional method of venous puncture. Variables related to children, intravenous therapy and professional characterization were collected. The dependent variables included the obtainment of peripheral venous access, the assertiveness, the catheter dwell time and the occurrence of local complications. For the statistical analysis were applied the Pearson Chi-square, Fisher's Exact, Generalization of Fisher's exact, Mann-Whitney, Likelihood Ratio and Prevalence Ratio (significance level of 5%).

ELIGIBILITY:
Inclusion Criteria:

* children submitted to intravenous therapy

Exclusion Criteria:

* adults

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 335 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Venous access obtainment occurred in the two studied groups, with marginally significant statistical difference. The success in the first attempt of puncture was statistically similar. | 1 year and 5 months

SECONDARY OUTCOMES:
The median of catheters dwell time was similar in the control group and experimental group. Infiltration had a different distribution between groups, been more frequent in the Experimental group. | 1 year and 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariane FM Avelar, Master, Principal Investigator — Federal University of São Paulo
Locations (1):
- São Paulo Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Avelar AF, Peterlini MA, da Pedreira ML. [Assertiveness and peripheral intravenous catheters dwell time with ultrasonography-guided insertion in children and adolescents]. Rev Esc Enferm USP. 2013 Jun;47(3):539-46. doi: 10.1590/s0080-623420130000300003. Portuguese. PMID 24601127